CLINICAL TRIAL: NCT04196725
Title: Effect of Lifestyle Intervention vs Physical Therapy Treatment in Patients With Secondary Lymphedema After Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: Montebellosenteret, Mesnali, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Montebello19
Record Dates: First submitted 2019-11-11; First posted 2019-12-12 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2019-12

CONDITIONS: Lymphedema, Secondary
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 26 participants will be enrolled in the cross over design consisting of two different rehabilitation programme. In addition there will be a parallel control group with 10 participants not participating in any of the rehabilitation programmes.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical therapy treatment (Experimental)
  Interventions: Other: Physical therapy treatment
- Lifestyle treatment (Experimental)
  Interventions: Behavioral: Lifestyle treatment
- Control (No Intervention): Parallel control group, not undertaking any treatment and not part of the cross-over design

INTERVENTIONS:
Other: Physical therapy treatment — Two weeks rehabilitation programme focusing on physical therapy treatment, e.g. manual lymphatic drainage and compression bandaging
  Arms: Physical therapy treatment
Behavioral: Lifestyle treatment — Two weeks rehabilitation programme focusing on physical activity
  Arms: Lifestyle treatment

SUMMARY:
Participants with lymphedema secondary to cancer treatment will participate in a two week rehabilitation programme focusing on physical therapy treatment and a two week programme focusing on physical exercise. The purpose is to assess the effect of the rehabilitation programmes on lymphedema and measures of physical performance.

DETAILED DESCRIPTION:
Traditionally, physical therapy treatment, e.g. manual lymphatic drainage and compression bandaging is used for treatment of cancer treatment induced lymphedema. Alternatively, lifestyle interventions are used as treatment, with focus on physical exercise. However, the effects of such interventions are scarcely documented. Thus, the purpose of this study is to assess the effect of physical therapy treatment and physical exercise on lymphedema and measures of physical performance.

The study will be performed in a randomized cross-over design, encompassing 26 participants with secondary lymphedema related to cancer treatment. Firstly, half of the participants in the intervention group will be randomized to a two week rehabilitation programme focusing on physical activity while the other half to a rehabilitation programme focusing on physical therapy treatment, and the other way around three months later. In addition. there will be a control group with cancer related lymphedema not participating in any rehabilitation programme. Pre and post of each of the two week rehabilitation periods the following measurements will be performed: The magnitude of lymphedema by volume measurements of the limbs (by DXA); measurements of maximal strength, range of movement, flexibility, balance, physical functionality and questionnaires about perceived health and level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Secondary lymphedema in arm or/and leg related to cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Lymphedema | Change from before to the end of each of the two week rehabilitation programmes.
  Ratio of the volume of affected limb vs volume of nonaffected limb measured by DXA

SECONDARY OUTCOMES:
Maximal strength | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  In handgrip and knee-extension
Balance | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  One leg balance test
Flexibility in hip and back | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  Sit and reach test
Flexibility in shoulder | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  Back scratch test
Test of physical functionality | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  Stand up and walk test
Range of joint movement in the knee, degrees of movement measured with a protractor | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  Range of joint movement in the knee
Range of joint movement in the elbow, degrees of movement measured with a protractor | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  Range of joint movement in the elbow
Self perceived health | Measured immediately before and at the end of each of the two week rehabilitation programmes.
  Perceived health assessed by questionnaire
Level of physical activity | Questionnaire will be completed immediately before the rehabilitation programmes, assessing the level of physical activity the prior three months.
  Level of physical activity assessed by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway